CLINICAL TRIAL: NCT01649336
Title: A Study of MEK162 and Paclitaxel in Patients With Epithelial Ovarian, Fallopian Tube or Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-162-112
Record Dates: First submitted 2012-07-22; First posted 2012-07-25 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — binimetinib; Paclitaxel; Antimitotic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MEK162 + paclitaxel (Experimental)
  Interventions: Drug: MEK162, MEK inhibitor; oral; Drug: Paclitaxel, mitotic inhibitor; intravenous

INTERVENTIONS:
Drug: MEK162, MEK inhibitor; oral — multiple dose, escalating
Drug: Paclitaxel, mitotic inhibitor; intravenous — multiple dose, single schedule

SUMMARY:
This is a Phase 1 study during which patients with platinum-resistant epithelial ovarian, fallopian tube or primary peritoneal cancer will receive investigational study drug MEK162 and paclitaxel. Patients will receive increasing doses of study drug in combination with paclitaxel in order to achieve the highest dose of study drug possible that will not cause unacceptable side effects. Patients will be followed to see what side effects the combination causes and what effectiveness the combination has, if any, in treating the cancer. Approximately 36 patients from the US will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of epithelial ovarian, fallopian tube or primary peritoneal cancer (measurable or evaluable, nonmeasurable disease) that is platinum-resistant or refractory. In the judgment of the Investigator, a patient who is platinum-sensitive but would not benefit from further platinum treatment is also eligible.
* Must have had ≥ 1 prior platinum-based chemotherapeutic regimen containing carboplatin, cisplatin or another organoplatinum compound for management of primary disease. This initial treatment may have included intraperitoneal (IP) therapy, consolidation, non-cytotoxic agents or extended therapy administered after surgical or non-surgical assessment.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2.
* Available archival tumor sample (excisional or core biopsy) that can be acquired and provide consent to biomarker testing of the tumor.
* Additional criteria exist.

Key Exclusion Criteria:

* History or concurrent evidence of retinal vein occlusion (RVO) or current risk factors for RVO.
* Prior therapy with a MEK inhibitor.
* History of hypersensitivity to taxanes or drug formulations containing Cremophor®.
* History of acute coronary syndromes.
* Uncontrolled or symptomatic brain metastases that are not stable, require steroids, are potentially life-threatening or that have required radiation within 28 days prior to first dose of study treatment.
* Concomitant malignancies or previous malignancies with less than a 5-year disease-free interval at the time of enrollment; patients with adequately resected basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or ductal carcinoma in situ may enroll irrespective of the time of diagnosis.
* Known positive serology for the human immunodeficiency virus (HIV), active hepatitis C, and/or active hepatitis B.
* Treatment with ritonavir at the time of first dose of study treatment.
* Treatment with continuous or intermittent small molecular therapeutics, biologic therapy or hormonal therapy within 28 days prior to first dose of study treatment.
* Treatment with a cyclical chemotherapy within a period of time that is less than the cycle length used for that treatment prior to first dose of study treatment.
* Treatment with any other investigational agents within a period of time that is less than the cycle length used for the treatment or within 28 days (whichever is shorter) prior to first dose of study treatment.
* Treatment with prior radiotherapy within 21 days prior to first dose of study treatment; however, if the radiation portal covered ≤ 10% of the bone marrow reserve, the patient may be enrolled irrespective of the end date of radiotherapy.
* Additional criteria exist.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Establish the recommended Phase 2 dose of study drug administered on continuous and intermittent schedules in combination with paclitaxel. | One year

SECONDARY OUTCOMES:
Characterize the safety profile of the study drug in combination with paclitaxel in terms of adverse events and clinical laboratory tests. | One year
Assess the efficacy of the study drug in combination with paclitaxel in terms of tumor response, duration of response and progression-free survival. | One year
Assess the potential plasma pharmacokinetic (PK) interactions between study drug, metabolites and paclitaxel in terms of plasma concentrations and noncompartmental PK parameters. | One year
Assess possible PK/efficacy and PK/safety correlations. | One year
Assess potential predictive biomarkers of clinical activity for the study drug in combination with paclitaxel. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Lafayette, Indiana
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Oklahoma City, Oklahoma